CLINICAL TRIAL: NCT01837550
Title: A Randomized, Controlled Trial Evaluating the Short- and Long-term Effects of an Internet-based Aural Rehabilitation Program for Hearing Aid Users Implemented in a General Clinical Practice
Brief Title: Educational Program for Hearing Aid Users With Internet Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sodra Alvsborgs Hospital (Other)
Responsible Party: Principal Investigator, Milijana Malmberg, PhD student, Principal Investigator, Sodra Alvsborgs Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HörNet VGR
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-03

CONDITIONS: Hearing Impaired
Keywords: audiologic rehabilitation; hearing loss; patient education; patient participation; structured rehabilitation; counseling; Internet
MeSH Terms: conditions — Hearing Loss; Patient Participation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): no professional support
  Interventions: Behavioral: Intervention group
- Intervention group (Experimental): Professional support via Internet
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Intervention group — The intervention group followed a five-week program that consisted of reading material, home training assignments, online and telephone interaction with an audiologist, and participation in a discussion forum.
  Arms: Control group
Behavioral: Control group — The control group only had access to reading material.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to examine the short-term effects of complementing an educational program for hearing aid users with Internet support.

DETAILED DESCRIPTION:
Aural rehabilitation aims to improve communication for people with hearing impairment. Education is widely regarded as an integral part of rehabilitation, but the effect of the delivery method of an educational program on the experience of hearing problems has rarely been investigated in controlled trials. Internet as a complement to aural rehabilitation has been tested in different studies with promising results. Though, until now not applied clinically as a part of an aural rehabilitation, focusing on hearing aid users with persistent self- reported hearing problems.

The purpose of this study was to evaluate the effect of an internet-based aural rehabilitation for hearing aid users from a clinical population.

Participants were randomly assigned to an intervention or control group. The intervention group followed a five-week program that consisted of reading material, home training assignments, online and telephone interaction with an audiologist, and participation in a discussion forum. The control group only had access to reading material.

The Hearing Handicap Inventory for the Elderly (HHIE), the Hospital Anxiety and Depression Scale (HADS) and the Communication Strategies Scale (CSS) were used to measure the outcomes of this study; and were recorded before and directly after the intervention as well as 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* the hearing aid users to be between 20 and 80 yr of age,
* the hearing aid users to have conductive or sensorineural hearing loss of mild to moderate degree (20-60 decibel Hearing Level pure-tone average measured across 500, 1000, and 2000 Hertz),
* the hearing aid users to have completed a hearing aid fitting at least 3 months before the study began (regardless of hearing aid manufacturer, model, or hearing aid outcomes),
* the hearing aid users to have a Hearing Handicap Inventory for the Elderly (HHIE) score of >20 points (indicative of some residual self-reported hearing problems),
* the hearing aid users to provide informed consent to participate

Exclusion Criteria:

* the hearing aid users who are not fulfilling the conditions to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Professor, Principal Investigator — Department of Clinical and Experimental Medicine, Division of Technical Audiology, Linkoping University, Sweden; Department of Behavioral Sciences and Learning, Swedish Institute.; Thomas Lunner, Professor, Principal Investigator — Department of Clinical and Experimental Medicine, Division of Technical Audiology, Linkoping University, Sweden; Oticon A/S, Research Centre Eriksholm, Snekkersten, Denmark.
Locations (1):
- Hearing Clinic, Hearing Organization, Borås, Vastra Gotalandsregion, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malmberg M, Lunner T, Kahari K, Andersson G. Evaluating the short-term and long-term effects of an internet-based aural rehabilitation programme for hearing aid users in general clinical practice: a randomised controlled trial. BMJ Open. 2017 Jun 6;7(5):e013047. doi: 10.1136/bmjopen-2016-013047. PMID 28592571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2013-2014; Borås Hospital, Sweden; Alingsås Hospital, Sweden; Skene Hospital, Sweden.
Pre-assignment Details: Participants who registered at the website and completed the screening form (n=108) were called for an interview to assess their eligibility; 104 informed an agreement to participate in the study. 14 of them did not fulfill the criteria for the Hearing Handicap Inventory for the Elderly, and 16 chose not to fill out the requested questionnaires.
Groups:
- Intervention Group: Professional support via Internet Intervention group: The intervention group is going to have access to a book and to a prepared compendium about communication strategies via the Internet and will receive weekly topic-based reading instructions related to the different chapters of the book or the compendium. The group will also have access to online and telephone support and access to an online discussion forum where new discussion topics will be posted each week. The project leader will evaluate the weekly data via the Internet.
- Control Group: no professional support
  Control group: The control group will only have access to the book's content via the Internet and will be asked to read and evaluate the content.
Period: T0-T1, 5 Weeks
Arm/Group | Intervention Group | Control Group
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0
Period: T0-T2, 6 Months Follow-up
Arm/Group | Intervention Group | Control Group
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (11.9) | 62.1 (11.4) | 62.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 24 | 20 | 44
Pure-tone average [Mean (Standard Deviation); unit: decibel Hearing Level] — Measuring the presence of conductive or sensorineural hearing loss of a mild to moderate degree, i.e., 20-60 dB HL. Pure-tone average (PTA) measured across 500-, 1000-, and 2000 Hz.
  decibel Hearing Level
    Right ear | 37.5 (11.3) | 38.0 (8.6) | 37.8 (10.0)
    Left ear | 37.8 (10.5) | 36.5 (8.5) | 37.1 (9.5)
Number of Hearing Aids [Number; unit: numbers]
  Binaurally | 28 | 31 | 59
  Monaurally | 9 | 6 | 15
Use of hearing aid [Mean (Standard Deviation); unit: years] | 7.5 (9.6) | 7.4 (6.3) | 7.5 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: The Hearing Handicap Inventory for the Elderly (HHIE)
Description: The HHIE measures the experience of hearing loss in older people by focusing on the psycosocial and emotional effects of hearing loss. Higher score reflects a higher self-reported hearing problem. Minimum score for the total scale (reported) is 0 and maximum score is 100 points.
Time Frame: 5 weeks, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 37 | 37
units on a scale
  Pre-measurement | 42.0 (16.9) | 36.1 (11.8)
  Directly after-measurement (5 weeks) | 35.8 (15.2) | 31.3 (14.3)
  6 months-post measurement | 36.0 (15.8) | 34.0 (13.2)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Non-Inferiority or Equivalence — To ensure a between-group effect of 80% at the 5% significance level it was estimated that 60 participants need to be included in the study. An effect size of Cohen's d=0.80 was expected. The expected standardized mean difference on the HHIE formed the basis for the obtained power; p = 0.685, Mixed Models Analysis

2. Secondary Outcome: International Outcome Inventory for Hearing Aids (IOI-HA)
Description: The IOI-HA measures hearing aid outcomes. The IOI-HA includes seven questions, measuring specific dimensions of hearing aid outcomes: daily use, benefits, remaining activity limitations, satisfaction, remaining participation restrictions, impact on the environment, and quality of life. Each question is scored from 1 to 5 (reported), where a higher score indicates a better outcome.
Time Frame: pre-measurement
Population: The IOI-HA was used only at the pre-masurement point, to select descriptive data about the participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 37 | 37
units on a scale
  1. Daily use | 4.1 (1.1) | 4.4 (1.0)
  2. Benefit | 3.8 (0.9) | 4.1 (0.9)
  3. Remaining activity limitation | 3.1 (0.8) | 3.1 (0.8)
  4. Satisfaction | 4.1 (1.1) | 4.4 (0.8)
  5. Remaining participation restriction | 3.8 (1.1) | 4.1 (0.8)
  6. Impact on environment | 3.6 (0.9) | 3.9 (0.9)
  7. Quality of life | 3.6 (0.8) | 3.6 (1.0)

3. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: The HADS contains 14 items. Responses are scored from 0 to 3 and a higher score indicates more symptoms of anxiety and depression. Minimum score for the total scale (reported) is 0 and maximum score for the total scale is 42.
Time Frame: 5 weeks, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 37 | 37
units on a scale
  Pre-measurement | 8.5 (6.6) | 7.4 (4.8)
  Directly after-measurement (5 weeks) | 7.5 (6.3) | 6.5 (5.2)
  6 months post-measurement | 4.8 (4.5) | 6.8 (5.9)

4. Secondary Outcome: Communication Strategies Scale (CSS)
Description: CSS is designed to analyze participants' behavior in various communication situations. Scoring for CSS ranges from 1 almost never to 5 almost always for subscales Verbal- and Nonverbal Strategies and conversely for Maladaptive Behaviors; indicating how frequent a specific situation or behavior occurs. Minimum score for the total scale (reported) is 0 and maximum score for the total scale is 125.
Time Frame: 5 weeks, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 37 | 37
units on a scale
  Pre-measurement | 68.1 (13.6) | 67.2 (11.3)
  Directly after-measurement (5 weeks) | 74.7 (11.1) | 68.5 (12.4)
  6 months post-measurement | 70.9 (10.5) | 66.7 (11.6)

ADVERSE EVENTS:
Time Frame: Directly after intervention (5 weeks), and 6 months post intervention
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No